CLINICAL TRIAL: NCT00937261
Title: Contrasting the Brain Effects of Risperidone and Invega With fMRI and PET Scanning
Brief Title: Contrasting the Brain Effects of Risperidone and Invega With Functional Magnetic Resonance Imaging (fMRI) and Positron Emission Tomography (PET) Scanning
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Irvine (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Steven G. Potkin, M.D., UC Irvine -FBIRN
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIRN 2008-6382
Record Dates: First submitted 2009-07-07; First posted 2009-07-10 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2010-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; Paliperidone Palmitate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Risperdal (Experimental): Risperdal 2-8mg per day
  Interventions: Drug: Risperidone
- Invega (Experimental): Invega 6-12mg per day
  Interventions: Drug: Paliperidone

INTERVENTIONS:
Drug: Risperidone — 2mg - 8mg per day, for the duration of participation in the study
  Other Names: Risperdal
  Arms: Risperdal
Drug: Paliperidone — 6mg - 12mg per day, for the duration of participation in the study
  Other Names: Invega
  Arms: Invega

SUMMARY:
The purpose of this study is to better understand brain function and psychiatric and neurological illness when taking Invega or Risperdal. The objective is to compare the brain effects of Invega to Risperdal in patients with Schizophrenia. This comparison will be evaluated with PET imaging, fMRI, and neurological ratings and assessments.

ELIGIBILITY:
Inclusion Criteria:

* are currently taking Risperdal and have been on the medication for at least three weeks
* are diagnosed with schizophrenia
* are able to provide written informed consent
* can safely have an MRI

Exclusion Criteria:

* are treatment resistant or intolerant to Risperdal
* have participated in another drug study in the past 28 days
* are pregnant or trying to become pregnant or are breastfeeding
* are colorblind
* have a history of alcohol, cannabis, or cocaine abuse within two weeks prior to the study
* have a current or past history of a major medical illness or have abnormal lab values which the study doctor feels is significant
* certain medications are also exclusionary including aripiprazole.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-07 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of BOLD signal activation and FDG metabolism of the DLPFC, superior temporal gyrus and amygdala, and their interaction between Invega and Risperdal | approximately 6-10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven G Potkin, M.D., Principal Investigator — UC Irvine
Locations (1):
- UC Irvine, Irvine, California, United States